CLINICAL TRIAL: NCT04131140
Title: Differences Across ICUs in Organ Donation After Brain Death: A Nationwide Study of Relationship With Variation in End-of-life Decisions
Brief Title: Organ Donation and End-of-life Decisions
Status: Completed | Type: Observational
Sponsor: Swedish Intensive Care Registry (Other)
Responsible Party: Sponsor
Other Study IDs: EPN2017/247-32
Record Dates: First submitted 2019-09-11; First posted 2019-10-18 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Decision Making; Terminal Illness; Tissue and Organ Procurement
Keywords: Advance Care Planning; Resuscitation Orders; Palliative Care; Brain Death; Organ Donation; Critical Illness; Intensive Care Units
MeSH Terms: conditions — Brain Death; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Variation in organ donation after brain death (DBD) per million population varies markedly between countries, within country regions, between and within intensive care units (ICU). These circumstances also apply to end-of-life decisions in the ICU.

The investigators studied all ICU deaths in Sweden between 2014-2017 in ICUs that, as routine, registered treatment plan (no treatment limitation and/or treatment limitation) and DBD.

The investigators hypothesized that ICUs with high proportion of treatment limitation (withholding or withdrawing life sustaining treatment) also had less proportion of DBD.

DETAILED DESCRIPTION:
The Swedish Intensive Care Registry (SIR) collects a comprehensive data set of patient characteristics, intensive care procedures, severity of illness scores, workload and outcomes using detailed guidelines.

Continuous data are collected as raw data, validated locally and transferred electronically to the registry for central validation (confirmed to be within prespecified limits and inconsistencies and illogical entries identified). If necessary, data are returned for correction and revalidation before being accepted and added to the master database. No data are changed by SIR. At SIR's homepage there are numerous open reports, updated as soon as new incoming data are processed by SIR.

SIR has an annual 2-day course for all ICU's in registration techniques and problems and daily telephone support possibilities concerning registration questions, problems and guidance. SIR has, however not yet a systematic on-site auditing program.

Missing data regarding treatment strategy are registered and are accounted for in the study. There are no missing data regarding organ donation.

The investigators calculate the proportion of treatment limitations per ICU as the number of deaths with any treatment limitation divided by all deaths in the same ICU.

Continuous variables are expressed as mean (standard deviations) or median (interquartile range).

Differences in proportions are analysed using the χ2-test. Changes over time are analysed using the non-parametric trend test. Survival are examined using the Kaplan-Meier estimate and differences in survival are analysed with the log-rank test.

Logistic regression is used to examine associations between patient and ICU characteristics and DBD as dependent variable. Mixed-effects logistic regression clustered per ICU is used to assess associations between treatment limitation and DBD after adjusting for patient age, sex, comorbidities, the Simplified Acute Physiology Score III (SAPS3) probability of death, principal diagnostic category, presence of treatment limitation and type of hospital.

Significance was assumed if P < 0.05.

ELIGIBILITY:
Inclusion Criteria:

All ICU deaths in Sweden between 1/1 2014 and 31/12 2017 from

1. general and neurological intensive care units,
2. which recorded treatment strategy according to national guidelines and
3. send data according to SIR's protocol for the follow-up of all deceased intensive care patients (DBD).

Exclusion Criteria:

1. Special units like paediatric (N=4), burn (N=2) and thoracic (N=8) intensive care units, due to low coverage ratio of documented treatment plan decisions in combination with a low ICU mortality rate.
2. General (N=3) ICUs that do not register documented treatment plan.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consisted of all ICU deaths (12,072) between 2014-2017 in general and neurological intensive care units which all recorded treatment strategy in their daily routine work.
  Special units like paediatric, burn and thoracic intensive care units were excluded
Sampling Method: Non-Probability Sample
Enrollment: 12072 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-03-22 (Actual)

PRIMARY OUTCOMES:
Rate of organ donations after brain death (DBD) | The estimated period of time to the ICU death is assessed up to 5 months after patient admission time to the ICU, with a median of 1.6 days. The event is determined by clinical examination or, in some cases cerebral angiography.
  Documented decision to carry out organ donation

SECONDARY OUTCOMES:
Rate of documented treatment limitations during ICU stay | The estimated period of time to the ICU documentation of treatment plan is assessed up to 5 months after patient admission time to the ICU, with a median of 14 hours. The event is determined by the note in patients medical record.
  Documented decision of treatment plan
Incidence and type of a documented treatment limitation during ICU stay | The estimated period of time to the ICU documentation of WH and/or WD medical treatment is assessed up to 5 months after patient admission time to the ICU, with a median of 14 hours. The event is determined by the note in patients medical record.
  Documented treatment plan is either 1) no treatment limitation or 2) treatment limitation, which then is specified as a) withholding (WH) and/or b) withdrawing (WD) of either mechanical ventilation (MV) and/or non-invasive ventilation (NIV) and/or continuous renal replacement therapy (CRRT) and/or vasoactive drugs.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas ÅI Nolin, MD, Study Director — The Swedish Intensive Care Registry (http://icuregswe.org); Nolin ÅI Thomas, MD, Principal Investigator — The Swedish Intensive Care Registry (http://icuregswe.org)
Locations (1):
- The Swedish Intensive Care Registry, Karlstad, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bendorf A, Kerridge IH, Stewart C. Intimacy or utility? Organ donation and the choice between palliation and ventilation. Crit Care. 2013 May 23;17(3):316. doi: 10.1186/cc12553. PMID 23714404
- [Background] Parker M, Shemie SD. Pro/con ethics debate: should mechanical ventilation be continued to allow for progression to brain death so that organs can be donated? Crit Care. 2002 Oct;6(5):399-402. doi: 10.1186/cc1542. Epub 2002 Aug 15. PMID 12398776
- [Background] Mark NM, Rayner SG, Lee NJ, Curtis JR. Global variability in withholding and withdrawal of life-sustaining treatment in the intensive care unit: a systematic review. Intensive Care Med. 2015 Sep;41(9):1572-85. doi: 10.1007/s00134-015-3810-5. Epub 2015 Apr 23. PMID 25904183
- [Background] Citerio G, Cypel M, Dobb GJ, Dominguez-Gil B, Frontera JA, Greer DM, Manara AR, Shemie SD, Smith M, Valenza F, Wijdicks EFM. Organ donation in adults: a critical care perspective. Intensive Care Med. 2016 Mar;42(3):305-315. doi: 10.1007/s00134-015-4191-5. Epub 2016 Jan 11. PMID 26754754
- [Background] Citerio G, Crippa IA, Bronco A, Vargiolu A, Smith M. Variability in brain death determination in europe: looking for a solution. Neurocrit Care. 2014 Dec;21(3):376-82. doi: 10.1007/s12028-014-9983-x. PMID 24865268
- [Background] Neitzke G, Rogge A, Lucking KM, Boll B, Burchardi H, Dannenberg K, Duttge G, Dutzmann J, Erchinger R, Gretenkort P, Hartog C, Jobges S, Knochel K, Liebig M, Meier S, Michalsen A, Michels G, Mohr M, Nauck F, Salomon F, Seidlein AH, Soffker G, Stopfkuchen H, Janssens U. [Decision-making support in Intensive Care to facilitate organ donation : Position paper of the Ethics Section and the Organ Donation and Transplantation Section of the German Interdisciplinary Association of Critical Care and Emergency Medicine (DIVI) in collaboration with the Ethics Section of the German Society of Medical Intensive Care Medicine and Emergency Medicine (DGIIN)]. Med Klin Intensivmed Notfmed. 2019 May;114(4):319-326. doi: 10.1007/s00063-019-0578-3. German. PMID 30976838
- [Background] Long AC, Brumback LC, Curtis JR, Avidan A, Baras M, De Robertis E, Efferen L, Engelberg RA, Kross EK, Michalsen A, Mularski RA, Sprung CL; Worldwide End-of-Life Practice for Patients in ICUs (WELPICUS) Investigators. Agreement With Consensus Statements on End-of-Life Care: A Description of Variability at the Level of the Provider, Hospital, and Country. Crit Care Med. 2019 Oct;47(10):1396-1401. doi: 10.1097/CCM.0000000000003922. PMID 31305497
- See also: Swedish Intensive Care Registry (SIR) is a national quality register for intensive care units. — http://www.icuregswe.org/
- See also: At the homepage of the Swedish Society for Anaesthesia and Intensive Care (SFAI) you find our national guidelines for treatment strategy in the intensive care units. English version at the link above. — https://sfai.se/wp-content/uploads/files/22-2%20Treatment_strategy.pdf
- See also: Sweden's national quality registries — http://www.kvalitetsregister.se/